CLINICAL TRIAL: NCT03181425
Title: Evaluation of Magnetic Resonance Imaging Diffusion Tensor and Knee Cartilage Tractography Reconstructions for the Study of Early Osteoarthritis
Brief Title: Magnetic Resonance Imaging Diffusion Tensor Tractography for Early Osteoarthritis Assessment
Acronym: TRACTILAGE
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Clinical Investigation Centre for Innovative Technology Network (Network)
Responsible Party: Sponsor
Other Study IDs: DCIC1614
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Knee Osteoarthritis
Keywords: Knee cartilage; Early Osteoarthritis; MRI tractography; Diffusion Tensor Imaging
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Imaging assessment: All subject of the study have a knee osteoarthritis (OA) and are going to have a knee prosthetic surgery with cartilage excision. Imaging measurements are conducted on human cartilage samples (2 samples per patient are selected : healthy and severely degraded).

SUMMARY:
The aim of this study is the evaluation of new MRI tractography maps for early knee osteoarthritis assessment.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is a common and chronic degenerative disease of the articular cartilage. Despite recent progress in the field of cartilage imaging, no routinely used clinical imaging modality has the ability to evaluate and monitor changes in cartilage degeneration.

More and more studies report the benefits of Magnetic Resonance (MR) diffusion tensor imaging (DTI) in the study of early knee osteoarthritis and in particular the new MRI contrasts generating the Track Weighted Imaging (TWI) technique.

This observationnal, pilot, prospective, unrandomized and uncontrolled study aim to evaluate, for the first time, the new MRI tractography maps for the assessment of early knee osteoarthritis. This study doesn't modify the medical care of the patient.

ELIGIBILITY:
Inclusion Criteria:

Over 18 years of age Knee prosthetic surgery indication with cartilage excision

Exclusion Criteria:

Refusal to sign a non-objection form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with knee arthoplasty indication
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of the MRI tractography reconstructions in the assessment of early osteoarthritis using the quantitative parameter of the average fiber lenght per voxel within a region of interest obtained from Average Pathlength Maps (APM). | 6 months
  Correlation between the average fiber lenght per voxel within a region of interest (APM maps) obtained from MRI tractography reconstructions of human cartilage and the gold standard of the arthrosis grade(OARSI).

SECONDARY OUTCOMES:
Evaluation of the MRI tractography reconstructions in the assessment of early osteoarthritis using a qualitative parameter of visual information obtained from APM maps. | 6 months
  Correlation between the qualitative parameter of visual information (heterogeneity, contrast density by fiber density) and the gold standard of the arthrosis grade(OARSI).
Evaluation the of the MRI tractography reconstructions in the assessment of early osteoarthritis using the Track Weighted - Apparent Diffusion Coefficient (TW-ADC) obtained from APM maps | 6 months
  Correlation between the Track Weighted - Apparent Diffusion Coefficient (TW-ADC) and the gold standard of arthrosis grade (OARSI).
Evaluation of MRI tractography reconstructions in the assessment of early osteoarthritis using the Track Weighted-Anisotropy Fraction (TW-FA) obtained from APM maps. | 6 months
  Correlation between the Track Weighted-Anisotropy Fraction (TW-FA) and the gold standard of arthrosis grade (OARSI).
Evaluation of MRI tractography reconstructions in the assessment of early osteoarthritis using the Track Weighted -Fibre Orientation Distribution (TW-FOD) obtained from APM maps. | 6 months
  Correlation between the Track Weighted -Fibre Orientation Distribution (TW-FOD) and the gold standard of arthrosis grade (OARSI).
Evaluation of MRI tractography reconstructions in the assessment of early osteoarthritis by using the Apparent Fibre Density (AFD) obtained from APM maps. | 6 months
  Correlation between the Apparent Fibre Density (AFD) and the gold standard of arthrosis grade (OARSI).
Evaluation of Optical Coherence Tomography (OCT) in the assessment of early osteoarthritis. | 6 months
  Correlation between the qualitative parameter from OCT and the gold standard of arthrosis grade (OARSI).
Sub-group analysis, according to the selected Anisotropy Fraction (FA) cutoff, to assess the MRI tractography reconstructions in the assessment of early osteoarthritis. | 6 months
  Correlation between the quantitative parameters previously cited and the gold standard of arthrosis grade (OARSI) for each group of Anisotropy Fraction (FA).

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Moreau-Gaudry, MD, PhD, Principal Investigator — Clinical Investigation Centre for Innovative Technology Network, University Hopital, Grenoble
Locations (1):
- Orthopedic Surgery Department, University Hopital Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Investigation Centre for Innovative Technology Network website — http://www.cic-it.fr/cic-it-grenoble.php